CLINICAL TRIAL: NCT01705977
Title: A Randomized, Double-Blind, Placebo-Controlled 52-Week Study to Assess Adverse Events of Special Interest in Adults With Active, Autoantibody-Positive Systemic Lupus Erythematosus Receiving Belimumab
Brief Title: Belimumab Assessment of Safety in SLE
Acronym: BASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115467; 2011-005667-25 (EudraCT Number); HGS1006-C1113 (Other: Human Genome Sciences Inc.)
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Antibodies; Lupus; SLE; Systemic Lupus Erythematosus; Autoimmune Disease; Belimumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — Standard of Care; belimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo plus standard therapy (Placebo Comparator): Placebo IV plus standard therapy; placebo administered on Days 0, 14, 28, and every 28 days thereafter through Week 48, with a final evaluation at Week 52 in the double-blind period.
  Interventions: Biological: Placebo plus standard therapy; Other: Standard therapy
- Belimumab 10 mg/kg plus standard therapy (Experimental): Belimumab 10 mg/kg IV plus standard therapy; belimumab administered on Days 0, 14, 28, and then every 28 days thereafter through Week 48, with a final evaluation at Week 52 in the double-blind period.
  Interventions: Biological: Belimumab 10 mg/kg plus standard therapy; Other: Standard therapy

INTERVENTIONS:
Biological: Placebo plus standard therapy — Placebo plus standard therapy
  Arms: Placebo plus standard therapy
Biological: Belimumab 10 mg/kg plus standard therapy — Belimumab 10 mg/kg plus standard therapy
  Other Names: BENLYSTA™
  Arms: Belimumab 10 mg/kg plus standard therapy
Other: Standard therapy — Standard therapy comprises any of the following (alone or in combination): corticosteroids, antimalarials, non-steroidal anti-inflammatory drugs (NSAIDs), and immunosuppressives; other biologics are not permitted.

SUMMARY:
The purpose of this study is to further enhance the existing knowledge regarding the side effects of belimumab when given with other lupus medicines to adults with active systemic lupus erythematosus (SLE). This study mainly focuses on collecting information on serious events that are not that common or may only be seen with long-term treatment. These events include death, serious infections and other infections of interest, cancers, serious mental health problems, including depression and suicide, and serious infusion and hypersensitivity reactions. This study is being done to help understand if treatment with belimumab increases the risk for these types of events. This study will also see if patients receiving belimumab with other lupus medicines can reduce their use of steroids, such as prednisone, over 1 year.

DETAILED DESCRIPTION:
Study participants receive standard therapy for SLE in addition to receiving the study drug, either placebo (no active medicine) or belimumab. The controlled period of the study is 52 weeks. The random assignment in this study is "1 to 1" which means that participants have an equal chance of receiving belimumab or placebo. After completion of the 52-week study period, participants will be contacted by phone annually for 4 more years to assess health status.

Following the 52-week controlled period, participants who wish to continue treatment with belimumab may be able to do so by being prescribed commercially available belimumab. If belimumab is not commercially available in the participant's country, the participant may be able to receive belimumab under a separate continuation protocol.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of SLE by American College of Rheumatology (ACR) criteria.
* Active SLE disease.
* Autoantibody-positive.
* On stable SLE treatment regimen which may include corticosteroids (for example, prednisone), antimalarial (for example, hydroxychloroquine) and/or immunosuppressants (for example, azathioprine, methotrexate, mycophenolate).

Key Exclusion Criteria:

* Pregnant or nursing.
* Have received treatment with any of the following: belimumab, either as a marketed product or as an investigational agent; any B cell targeted therapy (for example, rituximab) in the past year; or any biological agent (for example, adalimumab, etanercept, infliximab, or anakinra) in the past 90 days.
* Have received a live vaccine within the past 30 days.
* Have severe active lupus kidney disease.
* Have severe active central nervous system (CNS) lupus.
* Current or past positive for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4019 (Actual)
Dates: Start 2012-11-27 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (206):
- United States (44):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Covina, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Murrieta, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Cedar Rapids, Iowa
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, West Bloomfield, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Kalispell, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Hixson, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Cypress, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, McKinney, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Beckley, West Virginia
  - GSK Investigational Site, Clarksburg, West Virginia
- Argentina (13):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Lanús, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Zárate, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Venado Tuerto, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (4):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Fitzroy, Victoria
- Brazil (15):
  - GSK Investigational Site, Cuiabá, Mato Grosso
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Juiz de Fora, Minas Gerais
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Itajaí, Santa Catarina
  - GSK Investigational Site, São José do Rio Preto, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Campo Grande
  - GSK Investigational Site, Goiânia
  - GSK Investigational Site, Lajeado
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
- Bulgaria (8):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Shumen
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Targovisthe
  - GSK Investigational Site, Veliko Tarnovo
- Canada (2):
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Vaughan, Ontario
- Chile (2):
  - GSK Investigational Site, La Serena
  - GSK Investigational Site, Santigo
- Colombia (6):
  - GSK Investigational Site, Armenia
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Bucaramanga
  - GSK Investigational Site, Chía
  - GSK Investigational Site, Medellín
- Croatia (2):
  - GSK Investigational Site, Osijek
  - GSK Investigational Site, Rijeka
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Zlín
- GSK Investigational Site, Tallinn, Estonia
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Zalaegerszeg
- Indonesia (5):
  - GSK Investigational Site, Bandung
  - GSK Investigational Site, Denpasar
  - GSK Investigational Site, Malang
  - GSK Investigational Site, Palembang
  - GSK Investigational Site, Yogyakarta
- Italy (5):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Padua, Veneto
  - GSK Investigational Site, Pisa
- GSK Investigational Site, Klaipėda, Lithuania
- Malaysia (7):
  - GSK Investigational Site, Ipoh
  - GSK Investigational Site, Kota Bharu
  - GSK Investigational Site, Kota Kinabalu
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kuala Selangor
  - GSK Investigational Site, Kuala Terengganu
  - GSK Investigational Site, Seremban, Negeri Sembilan
- Mexico (10):
  - GSK Investigational Site, Torreón, Coahuila
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Cuautitlán Izcalli, State of Mexico
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, D.F
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, México
  - GSK Investigational Site, San Luis Potosí City
  - GSK Investigational Site, Torreón
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Wellington
- Peru (2):
  - GSK Investigational Site, Arequipa
  - GSK Investigational Site, Lima
- Philippines (7):
  - GSK Investigational Site, Angeles City, Pampanga
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Las Piñas
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Poland (3):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
- Portugal (5):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
  - GSK Investigational Site, Viseu
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Târgu Mureş
- Russia (6):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
- Serbia (4):
  - GSK Investigational Site, Belgrade
  - GSK Investigational Site, Kruševac
  - GSK Investigational Site, Niška Banja
  - GSK Investigational Site, Šabac
- GSK Investigational Site, Piešťany, Slovakia
- South Korea (7):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
- Spain (11):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Getafe/Madrid
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vilajoyosa
- Switzerland (2):
  - GSK Investigational Site, Sankt Gallen
  - GSK Investigational Site, Zurich
- Taiwan (5):
  - GSK Investigational Site, Chiayi County
  - GSK Investigational Site, Gueishan Township,Taoyuan County
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- Ukraine (12):
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Ternopil
  - GSK Investigational Site, Uzhhorod
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20766

REFERENCES:
- [Background] Sheikh S, Scheinberg MA, Wei CC, Tegzova D, Stohl W, Acayaba de Toledo R, Mucenic T, Abello M, Maksimowicz-McKinnon K, Abud Mendoza C, Navarra S, Garcia M, Garcia de la Torre I, Ordi Ros J, Nami A, Levy R, Bass D, Ross J, Punwaney R, Harris J, Pierce A, Thorneloe K, Ji B, Roth D. Mortality and adverse events of special interest in adult patients with active, auto-antibody-positive systemic lupus erythematosus receiving intravenous belimumab (BASE): a global, randomised, double-blind, placebo-controlled, multicentre Phase 4 trial. Lancet Rheumatol. 2020; DOI: 10.1016/S2665-9913(20)30355-6
- [Derived] Sheikh SZ, Scheinberg MA, Wei JC, Tegzova D, Stohl W, de Toledo RA, Mucenic T, Banfi MRA, Maksimowicz-McKinnon K, Abud-Mendoza C, Navarra S, Garcia M, Garcia-De La Torre I, Ros JO, Levy RA, Bass DL, Terres JR, Punwaney R, Harris J, Nami A, Pierce A, Thorneloe KS, Ji B, Roth DA. Mortality and adverse events of special interest with intravenous belimumab for adults with active, autoantibody-positive systemic lupus erythematosus (BASE): a multicentre, double-blind, randomised, placebo-controlled, phase 4 trial. Lancet Rheumatol. 2021 Feb;3(2):e122-e130. doi: 10.1016/S2665-9913(20)30355-6. Epub 2020 Dec 15. PMID 38279368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a global, multi-center, randomized, placebo-controlled double blind study that evaluated adverse events of special interest in adult participants with active, autoantibody-positive systemic lupus erythematosus (SLE) when treated with belimumab plus standard therapy versus participants who received placebo plus standard therapy for 1 year, followed by a Year 2-5 post-treatment follow-up period.
Pre-assignment Details: A total of 4019 participants were randomized in this study. 4003 participants who received at least one dose of study treatment contributed to the Intent-to-Treat (ITT) Population.
Groups:
- Placebo: Participants received placebo via the intravenous route on Days 0, 14, 28 and every 28 days through Week 48 with a final visit conducted at Week 52. Participants continued to receive standard SLE treatment and were followed up until end of study (up to 5 years).
- Belimumab 10 mg/kg: Participants received belimumab 10 milligrams per kilogram (mg/kg) on Days 0, 14, 28 and every 28 days through Week 48 with a final visit conducted at Week 52. Participants continued to receive standard SLE treatment and were followed up until end of study (up to 5 years).
Period: Treatment Period (Year 1)
Arm/Group | Placebo | Belimumab 10 mg/kg
Started | 2009 (Randomized) | 2010 (Randomized)
Intent-to-Treat Population | 2002 | 2001
Completed | 1729 | 1741
Not Completed | 280 | 269
Not completed — Withdrawal by Subject | 128 | 128
Not completed — Adverse Event | 57 | 49
Not completed — Protocol Violation | 2 | 4
Not completed — Site closure | 3 | 2
Not completed — Lost to Follow-up | 33 | 37
Not completed — Physician Decision | 48 | 38
Not completed — Missing study conclusion form | 2 | 2
Not completed — Randomized but not treated | 7 | 9
Period: Follow-up Period (Years 2 to 5)
Arm/Group | Placebo | Belimumab 10 mg/kg
Started | 1670 (1670 participants from the Year 1 - treatment period entered in the Year 2 to 5 follow-up period) | 1695 (1695 participants from the Year 1 - treatment period entered in the Year 2 to 5 follow-up period)
Completed | 1474 | 1514
Not Completed | 196 | 181
Not completed — Death | 58 | 38
Not completed — Lost to Follow-up | 75 | 89
Not completed — Withdrawal by Subject | 44 | 36
Not completed — Missing | 19 | 18

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for ITT Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Belimumab 10 mg/kg | Total
Number analyzed (Participants) | 2002 | 2001 | 4003
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (12.74) | 40.4 (12.75) | 40.6 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1853 | 1848 | 3701
  Male | 149 | 153 | 302
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian-European Heritage | 1070 | 1080 | 2150
  White/Caucasian-Arabic/North African Heritage | 19 | 16 | 35
  Mixed White Race | 1 | 0 | 1
  Asian-East Asian Heritage | 310 | 307 | 617
  Asian-South East Asian Heritage | 172 | 168 | 340
  Asian-Central/South Asian Heritage | 8 | 6 | 14
  Asian-Japanese Heritage | 2 | 1 | 3
  Mixed Asian Race | 0 | 1 | 1
  African American/African Heritage | 155 | 175 | 330
  Alaskan Native or American Indian | 257 | 228 | 485
  Native Hawaiian or Other Pacific Islander | 2 | 5 | 7
  Missing | 6 | 14 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Deaths - On Treatment Period (Week 52)
Description: Number of participants who died during on-treatment period (Week 52) is reported. The on-treatment period was defined as first dose to last dose + 28 days (or death). The As-Treated Population was defined as all participants who were randomized and received at least one dose of study agent,grouped according to the actual treatment administered for the majority (greater than [>]50 percent [%]) of the time. The on-treatment period was the primary analysis period for safety analyses.
Time Frame: Up to Week 52 (On-treatment period)
Population: As-Treated Population. One participant in placebo group who received belimumab >50% of the time was reported in the belimumab group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 2001 | 2002
Participants | 8 | 10
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.10, 95% CI 2-sided [-0.31 to 0.51] — 95% Confidence Interval was calculated using simple asymptotic Chi-Square (Pearson) method

2. Primary Outcome: Number of Participants Who Reported Protocol Defined Adverse Events of Special Interest (AESI): On-treatment Period (Week 52)
Description: A summary of protocol defined AESIs including serious infections, opportunistic infections and other infections of interest (serious and non-serious), non-melanoma skin cancer (NMSC), malignancies (excluding NMSC), psychiatric events suggesting serious mood disorders and anxiety (serious depression), suicidality (using Columbia-Suicide Severity Rating Scale [C-SSRS]) and serious infusion and hypersensitivity reactions (SIHR) is reported. The on-treatment period (Week 52) was defined as first dose to last dose + 28 days (or death). The on-treatment period was the primary analysis period for safety analyses.
Time Frame: Up to Week 52 (On-treatment period)
Population: As-Treated Population. One participant in placebo group who received belimumab >50% of the time was reported in the belimumab group. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 2001 | 2002
Participants
  Serious Infections, n=2001, 2002 | 82 | 75
  Opportunistic Infections and Other Infections of Interest, n=2001, 2002 | 50 | 36
  Malignancies (Excluding NMSC), n=2001, 2002 | 5 | 5
  NMSC, n=2001, 2002 | 3 | 4
  Psychiatric Events Suggesting Serious Mood Disorders and Anxiety (Serious depression), n=2001, 2002 | 1 | 7
  Suicidality (C-SSRS), n=1986, 1972: number analyzed (Participants) | 1986 | 1972
  Suicidality (C-SSRS), n=1986, 1972 | 23 | 28
  SIHR, n=2001, 2002 | 2 | 8
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = -0.35, 95% CI 2-sided [-1.55 to 0.85] — 95% CI for serious infections was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = -0.70, 95% CI 2-sided [-1.60 to 0.20] — 95% CI for opportunistic infections and other infections of interest (serious and non-serious) was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 3: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.00, 95% CI 2-sided [-0.31 to 0.31] — 95% CI for malignancies (excluding NMSC) was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 4: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.05, 95% CI 2-sided [-0.21 to 0.31] — 95% CI for NMSC was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 5: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.30, 95% CI 2-sided [0.02 to 0.58] — 95% CI for psychiatric events suggesting serious mood disorders and anxiety (serious depression) was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 6: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.26, 95% CI 2-sided [-0.44 to 0.96] — 95% CI for suicidality (C-SSRS) was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 7: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.30, 95% CI 2-sided [-0.01 to 0.61] — 95% CI for SIHR was calculated using simple asymptotic Chi-Square (Pearson) method

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Reported During On-treatment Period (Week 52)
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement. The on-treatment period (Week 52) was defined as first dose to last dose + 28 days (or death) and was the primary analysis period for safety analyses.
Time Frame: Up to Week 52 (On-treatment period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 2001 | 2002
Participants | 222 | 220

4. Secondary Outcome: Number of Deaths Reported - On-study Period (Week 52)
Description: Number of participants who died during on-study period (Week 52) is reported. The on-study period (which includes on and off treatment data) was defined as first dose to the end of the Week 52 study follow-up (or death). The on-study period was a supportive analysis period for safety analysis.
Time Frame: Up to Week 52 (On-study period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 2001 | 2002
Participants | 22 | 13
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = -0.45, 95% CI 2-sided [-1.03 to 0.13] — 95% CI was calculated using simple asymptotic Chi-Square (Pearson) method

5. Secondary Outcome: Number of Participants Who Reported Protocol Defined AESI: On-study Period (Week 52)
Description: A summary of protocol defined AESIs including serious infections, opportunistic infections and other infections of interest (serious and non-serious), NMSC, malignancies (excluding NMSC), psychiatric events suggesting serious mood disorders and anxiety (serious depression), suicidality (using C-SSRS) and SIHR is reported. The on-study period (Week 52) (which includes on and off treatment data) was defined as first dose to the end of the Week 52 study follow-up (or death). The on-study period was a supportive analysis period for safety analysis.
Time Frame: Up to Week 52 (On-study period)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 2001 | 2002
Participants
  Serious Infections, n=2001, 2002 | 95 | 80
  Opportunistic Infections and Other Infections of Interest, n=2001, 2002 | 59 | 39
  Malignancies (Excluding NMC), n=2001, 2002 | 7 | 5
  NMSC, n=2001, 2002 | 3 | 4
  Psychiatric Events Suggesting Serious Mood Disorders and Anxiety (Serious depression), n=2001, 2002 | 1 | 7
  Suicidality (C-SSRS), n=1988, 1974: number analyzed (Participants) | 1988 | 1974
  Suicidality (C-SSRS), n=1988, 1974 | 25 | 31
  SIHR, n=2001, 2002 | 2 | 8
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = -0.75, 95% CI 2-sided [-2.02 to 0.51] — 95% CI for serious infections was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 2: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = -1.00, 95% CI 2-sided [-1.96 to -0.04] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = -0.10, 95% CI 2-sided [-0.44 to 0.24] — 95% CI for malignancies (excluding NMSC) was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 4: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.05, 95% CI 2-sided [-0.21 to 0.31] — 95% CI for NMSC was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 5: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.30, 95% CI 2-sided [0.02 to 0.58] — [estimate comment as in outcome 2, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.31, 95% CI 2-sided [-0.42 to 1.05] — 95% CI for suicidality (C-SSRS) was calculated using simple asymptotic Chi-Square (Pearson) method
Statistical Analysis 7: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; Difference in percentage versus placebo = 0.30, 95% CI 2-sided [-0.01 to 0.61] — 95% CI for SIHR was calculated using simple asymptotic Chi-Square (Pearson) method

6. Secondary Outcome: Number of Participants With SAEs Reported During On-study Period (Week 52)
Description: A SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement. The on-study period (Week 52) (which includes on and off treatment data) was defined as first dose to the end of the Week 52 study follow-up (or death) and was a supportive analysis period for safety analyses.
Time Frame: Up to Week 52 (On-study period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 2001 | 2002
Participants | 241 | 233

7. Secondary Outcome: Percentage of Participants Whose Average Prednisone (or Equivalent) Dose to Treat SLE Has Been Reduced by >=25% From Baseline to <=7.5 mg/Day During Weeks 40 Through 52
Description: The average daily prednisone dose during Weeks 40 to 52 is the sum of all prednisone doses to treat SLE from the day following the Week 40 visit date up to but not including the Week 52 study completion date divided by the number of days between Week 40 visit date and study completion date (study completion date - Week 40 visit date). Percentage of participants whose average prednisone dose has been reduced by >=25% from Baseline to <=7.5 mg/day during Weeks 40 through 52 in participants with average prednisone use greater than 7.5 mg/day at Baseline was compared between belimumab and placebo using a logistic regression model including treatment group, Baseline prednisone dose, screening safety of estrogen in lupus national assessment (SELENA) systemic lupus erythematosus disease activity index (SLEDAI) score (<=9 versus >=10) and region. Baseline is defined as the last available value measured prior to dosing on or before the date of first dose (Day 1).
Time Frame: Week 40 to Week 52
Population: ITT Population. Only those participants with Baseline prednisone>7.5 mg/day were analyzed. The ITT population is defined as all participants who were randomized and received at least one dose of study agent and the analysis was performed per the treatment that a participant was randomized to receive, regardless of the actual treatment received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 990 | 986
Percentage of Participants | 16.2 | 19.9
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; p = 0.0284, Regression, Logistic; Odds ratio versus placebo = 1.30, 95% CI 2-sided [1.03 to 1.65] — 95% CI and P-value was calculated from a logistic regression model for the comparison between belimumab and placebo including treatment group, Baseline prednisone dose, screening SELENA SLEDAI score (<=9 versus >=10) and region

8. Secondary Outcome: Number of Participants With All-cause Mortality During Years 2 to 5
Description: Number of participants with all-cause mortality during years 2 to 5 has been presented.
Time Frame: From 2 years to 5 years
Population: As-Treated Any Year 2-5 Follow-up Population consisted of all participants in the As-Treated population who completed at least one post-treatment follow-up visit for Year 2 to 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 1670 | 1695
Participants | 58 | 38

9. Secondary Outcome: Number of Participants With New Primary Malignancies During Years 2 to 5
Description: Number of participants with new primary malignancies during years 2 to 5 has been presented.
Time Frame: From 2 years to 5 years
Population: As-Treated Any Year 2-5 Follow-up Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 1670 | 1695
Participants | 22 | 24

ADVERSE EVENTS:
Time Frame: AESIs and all SAEs were collected up to Week 52 (On-study period), all-cause mortality was collected up to end of study (up to 5 years)
Description: All-cause mortality, AESIs and SAEs are summarized for the As-Treated Population. Only AESIs and SAEs were collected up to Week 52, but not all AEs. All-cause mortality was collected up to end of study (up to 5 years). One participant in placebo group who received belimumab >50% of the time was reported in the belimumab group
Arm/Group | Placebo | Belimumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 80/2001 | 51/2002
Serious Adverse Events (participants affected / at risk) | 241/2001 | 233/2002
Other Adverse Events (participants affected / at risk) | 31/2001 | 17/2002
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2001) | Belimumab 10 mg/kg (N=2002)
Pneumonia (Infections and infestations) | 27 (28) | 18 (18)
Urinary tract infection (Infections and infestations) | 8 (9) | 16 (17)
Lupus nephritis (Renal and urinary disorders) | 11 (11) | 6 (6)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 11 (12) | 5 (6)
Cellulitis (Infections and infestations) | 8 (8) | 7 (7)
Gastroenteritis (Infections and infestations) | 11 (11) | 4 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 2 (2)
Pyrexia (General disorders) | 6 (6) | 2 (2)
Sepsis (Infections and infestations) | 4 (5) | 4 (4)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 6 (6)
Septic shock (Infections and infestations) | 3 (3) | 4 (4)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Herpes zoster (Infections and infestations) | 5 (5) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 1 (2)
Appendicitis (Infections and infestations) | 2 (2) | 3 (3)
Pulmonary tuberculosis (Infections and infestations) | 4 (4) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 3 (3)
Suicide attempt (Psychiatric disorders) | 1 (1) | 4 (4)
Urosepsis (Infections and infestations) | 2 (2) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 3 (4)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Ovarian cyst (Reproductive system and breast disorders) | 1 (2) | 3 (3)
SLE arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 3 (3)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 1 (1)
Central nervous system vasculitis (Nervous system disorders) | 1 (1) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 3 (3) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 2 (2)
Endometriosis (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dengue haemorrhagic fever (Infections and infestations) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Encephalitis (Infections and infestations) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 2 (2)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lupus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lupus vasculitis (Vascular disorders) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Superinfection (Infections and infestations) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Uterine haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anomalous pulmonary venous connection (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bartholinitis (Infections and infestations) | 0 (0) | 1 (1)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system lupus (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus mucocutaneous ulcer (Infections and infestations) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hookworm infection (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Jaundice extrahepatic obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Joint tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lupus enteritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Lupus pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis listeria (Infections and infestations) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (2)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Neuropsychiatric lupus (Nervous system disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema due to renal disease (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adhesion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ovulation pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periorbital swelling (Eye disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Serositis (General disorders) | 0 (0) | 1 (1)
Shrinking lung syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis gastrointestinal (Infections and infestations) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vasculitis necrotising (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2001) | Belimumab 10 mg/kg (N=2002)
Herpes zoster (Infections and infestations) | 31 (33) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT01705977/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT01705977/SAP_003.pdf